CLINICAL TRIAL: NCT05334901
Title: Effect of Different Curing Times and Intensities on The Performance of Compound Class II Bulk-Fill Resin Composite Restorations: (An In-Vivo and In-Vitro Study)
Brief Title: Performance of Curing Times and Intensitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Roaa Sabry, roaa.sabry@dentistry.cu.edu.eg, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPR 22/3/2022
Record Dates: First submitted 2022-03-22; First posted 2022-04-19 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Clinical Performance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High intensity light cure (Experimental): High intensity light curing (2200 mw/cm2)To achieve increased power and a wider spectrum for short exposure time (1 second) to overcome resin composite restoration techniques sensitivity and shorten the clinical procedure
  Interventions: Device: High intensity light cure
- Low intensity light cure (Active Comparator): Conventional light curing (1200 mw/cm2) for long exposure time (20 seconds) to achieve the slower rate of conversion allowing for a better flow of the material, which decreases contraction stress in the filling material
  Interventions: Device: High intensity light cure

INTERVENTIONS:
Device: High intensity light cure — Bulk fill resin composite restoration cured with high intensity light curing (2200 mw/cm2)To achieve increased power and a wider spectrum for short exposure time (1 second) to overcome resin composite restoration techniques sensitivity and shorten the clinical procedure

SUMMARY:
The aim of the study is to compare the effect of high intensity light cure (2200 mw/cm2) for 1 second with low intensity light cure (1200 mw/cm2) for 20 seconds on the clinical performance of bulk fill resin composite restorations in compound Class II cavities of posterior teeth

DETAILED DESCRIPTION:
The prepared cavities will be conditioned with 35% phosphoric acid gel for15 seconds, then will be rinsed and dried with compressed air. Then application of universal adhesive system to all cavity with bond brush then light cured for 10 seconds using LED light curing unit (1200 mw/cm2). Extra-Fill bulk fill resin composite will be applied in onebulk increment and will be light polymerized for 1 second using (LED) light curing unit (2200 mw/cm2).for intervention group Extra-Fill bulk fill resin composite will be applied in one bulk increment and will be light polymerized for 20 seconds using (LED) light curing unit (1200 mw/cm2) fot control group

ELIGIBILITY:
Inclusion Criteria:

* Permanent premolars or molars.
* Moderate to deep compound class II cavities.
* Vital with the positive reaction to a cold thermal stimulus.
* Absence of parafunctional habits

Exclusion Criteria:

* Teeth with clinical symptoms of pulpitis such as spontaneous pain or sensitivity to pressure.
* Non-vital teeth.
* Secondary carious lesions.
* Advanced periodontal disease

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Clinical performance | Change from the baseline at 6 months and12 months
  Clinical performance of bulk fill resin composite restorations will be evaluated by modified USPHS Criteria includes:
  * Marginal Discoloration
  * Marginal adaptation
  * Secondary caries
  * Postoperative sensitivity
  For each criteria one score will be chosen from 3 scores (Alpha,Bravo&Charlie).

CONTACTS AND LOCATIONS:
Overall Officials: Roaa Azazy, Master, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry, Giza, Cairo Governorate
  - Faculty of Dentistry, Cairo

IPD SHARING:
Plan to Share IPD: Yes
The aim of the study is to compare the effect of high intensity light cure (2200 mw/cm2) for 1 second with low intensity light cure (1200 mw/cm2) for 20 seconds on the clinical performance of bulk fill resin composite restorations incompound Class II cavities of posterior teeth
Supporting Information: Study Protocol
Time Frame: T0: baseline (after one week) T1: after 6 months T2: after 12 months
Access Criteria: 1. Permanent premolars or molars.
  2. Moderate to deep compound class II cavities.